CLINICAL TRIAL: NCT06056752
Title: A Dose-escalation Clinical Study of QH103 Cell Injection (CD19 CAR-γδT Cell Injection) in Patients With Relapsed/Refractory B-cell Acute Lymphoblastic Leukemia (B-ALL).
Brief Title: QH103 Cell Injection for the Treatment of Relapsed/Refractory B-cell Acute Lymphoblastic Leukemia
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Anhui Provincial Hospital (Other Government)
Responsible Party: Principal Investigator, Xiaoyu Zhu, Director of Hematology Department, Anhui Provincial Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: QH10302-B-01(0)
Record Dates: First submitted 2023-09-21; First posted 2023-09-28 (Actual); Last update posted 2023-10-24 (Actual); Status verified 2023-10

CONDITIONS: B-cell Acute Lymphoblastic Leukemia
Keywords: B-ALL; Allogenic CAR-γδT Cell; CD19; cell therapy
MeSH Terms: conditions — Burkitt Lymphoma | interventions — fludarabine; fludarabine phosphate; Injections; Cyclophosphamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients with relapsed/refractory CD19-positive B-cell acute lymphoblastic leukemia (Experimental): A conditional chemotherapy regimen of fludarabine and cyclophosphamide will be administered, followed by investigational therapy, QH103 Cells
  Interventions: Biological: QH103 Cell Injection; Drug: Fludarabine; Drug: Cyclophosphamide

INTERVENTIONS:
Biological: QH103 Cell Injection — dose escalation (3+3) : dose 1 (3×10^8CAR+cells) ,dose 2 (1 × 10^9 CAR+cells）,dose 3 (3 × 10^9CAR+cells)
Drug: Fludarabine — Intravenous fludarabine on days-5~-2,the infusion dose is adjusted according to the subject's condition
  Other Names: Fludarabine Phosphate for Injection
Drug: Cyclophosphamide — Intravenous cyclophosphamide on days -5~-3, the infusion dose is adjusted according to the subject's condition
  Other Names: Cyclophosphamide for Injection

SUMMARY:
This is a single-arm, single-center, interventional, dose-escalation clinical study designed to evaluate the safety and tolerability of QH103 Cell Injection in the treatment of patients with relapsed/refractory B-cell acute lymphoblastic leukemia.

DETAILED DESCRIPTION:
To evaluate the safety and tolerability of QH103 Cell Injection in the treatment of relapsed/refractory CD19-positive B-cell acute lymphoblastic leukemia, and to evaluate dose-limiting toxicity and maximum tolerated dose.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥14 years, gender is not limited;
2. Patients with clinically diagnosed relapsed/refractory B-ALL (except those presenting with extramedullary disease only), including any of the following:

   1. Failure to obtain CR after 2 cycles of standard chemotherapy;
   2. First induction of CR, but duration of CR is ≤12 months;
   3. Relapsed/refractory B-ALL that has failed to respond to the first or multiple salvage treatments;
   4. Relapse after hematopoietic stem cell transplantation, including hematological relapse and positive micro residual disease (MRD).
3. Cytological or histological confirmation of tumor cell immunophenotyping as CD19 positive;
4. Bone marrow with a ratio of ≥5% primitive/naïve lymphocytes (morphology);
5. Expected survival time of more than 3 months;
6. Eastern Cooperative Oncology Group (ECOG) score of 0-2;
7. Vital organ function meets the following requirements: left ventricular ejection fraction ≥50% on echocardiography; serum creatinine≤1.5 × upper limit of normal range (ULN); glutamine aminotransferase, aspartate aminotransferase ≤3 times ULN, total bilirubin ≤1.5 times ULN;
8. Pregnancy tests for women of childbearing age should be negative, and both men and women should agree to use effective contraception during treatment and for the following 1 year.
9. Toxicity of prior antitumor therapy ≤ grade 1 (according to CTCAE version 5.0) or acceptable inclusion/exclusion criteria level.
10. No significant hereditary disease;
11. Be able to understand the requirements and matters of the trial and be willing to participate in the clinical study as required;
12. Sign the trial informed consent form.

Exclusion Criteria:

1. with uncontrolled active central nervous system leukemia (CNSL) or a history of epilepsy, cerebrovascular disease
2. Pregnant or lactating women, or those who do not consent to the use of the drug during and within 1 year after treatment;
3. Other malignant tumors not in remission;
4. with primary immunodeficiency or autoimmune diseases requiring immunosuppressive therapy;
5. Patients who have received immune cell therapy within 6 months prior to enrollment and donor lymphocyte infusion within 6 weeks prior to enrollment.
6. Patients with confirmed positive serum anti-FMC63 and DSA reactions;
7. Patients who have participated in other clinical trials within 4 weeks prior to enrollment;
8. Uncontrolled infectious or other serious diseases, including but not limited to infections (Human Immunodeficiency Virus, acute or chronic active hepatitis B or hepatitis C), congestive heart failure, unstable angina pectoris cardiac arrhythmias, or conditions that the attending physician considers to be an unpredictable risk;
9. Uncontrollable plasma fluid, such as large pleural effusions or ascites;
10. History of stroke or intracranial hemorrhage within 3 months prior to enrollment;
11. Major surgery or trauma within 28 days prior to enrollment, or major side effects from which you have not recovered;
12. History of allergy to any of the ingredients in the cellular product;
13. Inability to understand or unwillingness to sign the informed consent form;
14. Other reasons deemed by the investigator to be unsuitable for the clinical trial.

Min Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2023-09-27 (Actual); Primary Completion 2025-07-03 (Estimated); Study Completion 2026-07-03 (Estimated)

PRIMARY OUTCOMES:
Incidence of Adverse Events (AEs) | 12 months
  AE is defined as any adverse medical event from the date of leukapheresis to 12 months after QH103 infusion. Among them, cytokine release syndrome (CRS) and immune cell-associated neurotoxicity syndrome (ICANS) were graded according to American Society for Transplantation and Cellular Therapy (ASTCT) criteria, graft-versushost disease (GVHD) according to criteria defined by the Mount Sinai Acute GVHD International Consortium. Other AEs were graded according to common terminology criteria for adverse events (CTCAE) v5.0
Incidence of Dose-Limiting Toxicities (DLTs) | First infusion date of QH103 cells to 28 days end cell infusion
  DLT was defined as QH103 Cells-related events with onset within first 28 days following infusion:
  The development of Grade (G) III-IV acute GVHD according to the Mount Sinai Acute GVHD International Consortium criteria; The development of G3 or higher grade CRS lasting > 2 weeks; Any QH103 cells-related AE requiring intubation; All G4 non-hematologic toxicities. Symptoms of GVHD include but are not limited to skin rash, enterocolitis with diarrhea, liver dysfunction with jaundice, fever, weight loss, etc.
Maximum tolerated dose (MTD) | 28 days
  MTD is defined as the highest dose level of less than or equal to 2 DLT among the 6 subjects finally determined.

SECONDARY OUTCOMES:
Overall Survival (OS） | 12 months
  OS is defined as the time from QH103 cells infusion to the date of death. Subjects who have not died by the analysis data cutoff date will be censored at their last contact date.
Progression Free Survival (PFS) | 12 months
  PFS is defined as the time from the QH103 cells infusion date to the date of disease progression assessed by investigators assessment, or death any cause. Participants not meeting the criteria for progression by the analysis data cutoff date were censored at their last evaluable disease assessment date.
Pharmacokinetics: Persistence of the QH103 cells | 28 days
  Persistence of the QH103 cells assessed by number in peripheral blood.
Pharmacodynamics: Peak level of cytokines in serum | 28 days
  The cytokines mainly include interleukin-2 (IL-2 ), IL-6, IL-8, IL-10, tumor necrosis factor-α (TNF-α) etc. Peak was defined as the maximum post-baseline level of the cytokine.
Overall Response Rate(ORR) | 12 months
  Proportion of subjects with CR (complete response) and CRi (complete response with incomplete hemocyte recovery)

CONTACTS AND LOCATIONS:
Overall Officials: Xiaoyu Zhu, Ph.D, Principal Investigator — Director of Hematology Department, Anhui Provincial Hospital
Locations (1):
- Anhui Provincial Hospital, Hefei, Anhui, China